CLINICAL TRIAL: NCT06483867
Title: A Study of the Correlation Between NIRS Monitoring Early Postnatal Tissue Oxygen Saturation and Clinical Outcomes in Very Preterm Infants: A Single-center Prospective Cohort Study
Brief Title: The Correlation Between Tissue Oxygenations Using NIRS and Clinical Outcomes in Very Preterm Infants.
Acronym: TCBTOUNACOIVPI
Status: Not yet recruiting | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: huiwu
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-02

CONDITIONS: Tissue Oxygenation
Keywords: Very preterm infants; composite outcome; Near-Infrared Spectroscopy; Tissue oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With the development of neonatal critical medicine, the survival rate of premature infants has gradually increased, and the incidence of late complications has significantly decreased, but preterm delivery is still the main cause of death of children in China.

Near infrared spectroscopy (NIRS) makes use of the different absorption spectra of oxygenated and deoxyhemoglobin in the near infrared band to provide tissue oxygenation index, which is non-invasive and convenient. Due to the thin skin and bone of newborns, near infrared spectroscopy has a broad prospect and important significance in the field of newborns. Non-invasive, real-time and continuous monitoring of brain oxygenation, intestinal oxygenation and tissue perfusion of premature infants can provide doctors with important information support and auxiliary means, which can help to detect and deal with various complications in time and improve the survival rate and health status of premature infants. The current research is mainly focused on exploring the relationship between some specific indicators and corresponding diseases, but there is a lack of research on a series of complications related to premature infants, especially in very premature infants, due to the immaturity of multiple organ system development. They had a significantly higher risk of complications such as severe intraventricular hemorrhage, necrotizing enterocolitis (NEC), retinopathy of prematurity (ROP), bronchopulmonary dysplasia (BPD) and so on. However, there is a lack of cohort study on the prediction of early complications in such children. The purpose of this study is to further explore the changes of tissue oxygen saturation and related indexes in the early postnatal period and their relationship with related complications. It is assumed that the tissue oxygen saturation in the early postnatal period is related to the adverse outcome in hospital, so as to intervene the children early and reduce the occurrence of adverse outcome.

DETAILED DESCRIPTION:
NIRS monitoring begins within 24 hours after birth. Oxygen saturation in the brain and intestines is monitored for 15 minutes at the same time every day. The probe should be fixed with medical tape and closed to the skin to avoid light leakage. At the same time, shading measures should be taken on the probe and skin surface to reduce the impact of environmental factors. Continuous monitoring for 7 days. If the infants start feeding during the period, monitor 15 minutes from 5 minutes before feeding, including before, during, and after feeding, and the relatively stable data at each time point was taken as the intestinal tissue oxygen saturation at that time, and the oxygen saturation variation and tissue oxygen extraction ratio are calculated. Clinical data were recorded at the time of each measurement and included feeding status and the use of mechanical ventilation, oxygen therapy, and medications and so on.

ELIGIBILITY:
Inclusion Criteria:

* (1) All infants born at <32 weeks of gestation. (2) Register and start NIRS monitoring within 24 hours after birth; (3) Obtain the written consent of parents.

Exclusion Criteria:

* Potential sensor interference: Disorders of/nonkeratinized skin; Hydrops/anasarca; Severe jaundice; Chromosomal abnormality ；Severe congenital malformations； Parents refuse to participate

Ages: 0 Hours to 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: (1) All infants born at <32 weeks of gestation. (2) Register and start NIRS monitoring within 24 hours after birth; (3) Obtain the written consent of parents.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
The composite outcome | 2023.12-2024.12
  death or any 1 of the following morbidities: bronchopulmonary dysplasia (BPD), retinopathy of prematurity ≥stage 3,periventricular leukomalacia, Necrotizing Enterocolitis≥stage II, and sepsis